CLINICAL TRIAL: NCT06891092
Title: Comparison of Quality of Vision After Implantation of Monofocal Depth-enhanced Intraocular Lenses in Patients Undergoing Bilateral Cataract Surgery
Brief Title: Vivinex Impress XY1-EM vs RayOne EMV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1778
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cataract
Keywords: non-diffractive monofocal IOL; EDOF; cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rayone EMV (Experimental): Patient will receive the non-diffractive monofocal IOL during cataract surgery
  Interventions: Device: RayOne EMV
- Vivinex Impress XY1-EM (Experimental): Patient will receive the non-diffractive monofocal IOL during cataract surgery
  Interventions: Device: Vivinex Impress

INTERVENTIONS:
Device: RayOne EMV — non-diffractive monofocal IOL
  Arms: Rayone EMV
Device: Vivinex Impress — non-diffractive monofocal IOL
  Arms: Vivinex Impress XY1-EM

SUMMARY:
Comparison of the outcomes of bilateral implantation of extended depth of vision (EDOF) intraocular lenses (IOLs): the Rayone EMV and the Vivinex Impress XY1-EM in patients with cataract

DETAILED DESCRIPTION:
Cataracts are one of the leading causes of visual impairment and blindness worldwide. Modern cataract surgery by phacoemulsification with intraocular lens implantation is the gold standard of treatment. Conventional monofocal intraocular lenses are still the most commonly used intraocular lenses today. They allow good uncorrected visual acuity to the far distance, while the patient can achieve good visual acuity to the intermediate near distance with glasses.

However, in developed countries, patients expect good quality vision not only to the far distance, but also to intermediate and near distances due to the many daily activities that require this range of vision (reading on tablets and smartphones, driving, carrying on a conversation). To meet these expectations, most intraocular lens manufacturers have introduced extended depth-of-field lens technology, which provides good visual acuity for distance and intermediate distances with few visual side effects. These lenses achieve satisfactory uncorrected visual acuity not only for distance, but also for near and intermediate distances.

Summarising the above arguments, it therefore seems that implanting patients with lenses that allow good distance vision and satisfactory vision to intermediate and near distances can result in an increased quality of life after cataract surgery.

Characteristics of the lenses tested RayOne EMV RAO200E lens (Rayner Intraocular Lenses Ltd) -This lens was developed in collaboration with Professor Graham Barrett. It is a preloaded monofocal+/non-diffractive EDOF, hydrophilic lens that provides an extended range of vision by exploiting positive spherical aberration. The overall diameter of the lens is 12.5mm and the optical diameter is 6.0mm. The lens has an aspherical front surface, biconvex shape. Its effect is to amplify/compensate for the cornea's natural positive spherical aberration, resulting in an increased range of acuity. As it meets ISO standards for monofocal intraocular lenses, it is less affected by variable pupil width, decentration and tilt. The RayOne EMV can be used for bilateral emmetropia and is also optimised for use in a monovision system. For emmetropia, it allows better intermediate vision than standard monovision lenses, providing approximately 1.25 D of extended visual range Vivinex impress XY1-EM (Hoya Surgical Optics, Singapore) - is a new monofocal lens made of hydrophobic non-gloss acrylate with aspheric optics that provides extended depth of field in the intermediate range. It has a combination of standard aspheric and even aspheric surface with microscopic angles. No first studies on the clinical properties of this enhanced monofocal lens are available in the literature.

From the available literature, it appears that both lenses have similar visual improvement efficacy with a similar safety profile. There is currently no study in the available literature directly comparing the two in a randomised manner.

The prospective randomised study will encompass 100 eyes of patients at the Department of Ophthalmology, Medical University of Bialystok, suffering from cataracts in both eyes, qualified for surgical treatment by simultaneous phacoemulsification in both eyes on one day between 2025 and 2028. This method is widely used worldwide. In the local clinic, it was introduced during the Covid-19 pandemic, when hospital visits had to be reduced due to epidemiological risks and the need for social distancing. At present, about 15% of all cataract operations at the clinic here are simultaneous bilateral procedures. Patients who have had no previous ophthalmic surgery and whose health status allows them to participate in the study within 3 months will be eligible. Randomisation will be performed on the day of the patient's qualification for the surgery by means of a draw of the type of lens written on a card placed in a closed envelope.

Group I patients (n=50) will be implanted with Vivinex Impress XY1-EM lenses, group II with RayOne EMV lenses (n=50). Qualification for binaural cataract surgery will be according to NHF guidelines: visual acuity <60% of normal.

Operations will be performed by several, experienced operators. Patients' quality of vision will be assessed 2 times: before surgery and 3 months after surgery using the Visual Function Index Questionnaire (VF 14). The VF-14 is a short questionnaire designed to measure functional motor impairment in cataract patients. It consists of 18 questions covering 14 aspects of visual function of cataract patients. The VF-14 demonstrates high internal consistency and is reliable, providing information that cannot be conveyed by measures of visual acuity or general health. The experiment will be discontinued if the above lenses are found to have an adverse effect on patients' visual quality or biological side effects are identified.

ELIGIBILITY:
Inclusion Criteria:

* age-related bilateral cataract
* age 21 or older
* visual acuity > 0.05
* axial length: 22.0 - 26.0 mm
* normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* written informed consent prior to surgery

Exclusion Criteria:

* active ocular disease (e.g. chronic severe uveitis, proliferative diabetic retinopathy, chronic glaucoma not responsive to medication)
* relevant other ophthalmic diseases such as pseudoexfoliation syndrome (PEX), intraoperative floppy iris syndrome (IFIS)
* corneal decompensation or corneal endothelial cell insufficiency
* previous ocular surgery or trauma
* persons who are pregnant or nursing (pregnancy test will be taken in women of reproductive age)
* corneal astigmatism > 1 dpt.
* retinopathies

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity at intermediate distance | 3 months
  The visual acuity at the intermediate distance will be measured using ETDRS charts at a distance of 80 centimetres and compared between the two different IOLs. The higer the number the better outcome.

SECONDARY OUTCOMES:
Visual acuity at far distance | 3 months
  The visual acuity at the far distance will be measured using ETDRS charts at a distance of 4 metres and compared between the two different IOLs. The higer the number the better outcome.
Visual acuity at near distance | 3 months
  The visual acuity at the near distance will be measured using ETDRS charts at a distance of 40 centimetres and compared between the two different IOLs. The higer the number the better outcome.
Change from baseline in the quality of life | 3 months
  Patients' quality of vision will be measured with the Visual Function Index Questionnaire and compared to outcome prior surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Bialystok, Bialystok, Polska, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data that underlie the results reported in this study will be available upon reasonable request for academic and non-commercial purposes beginning with results publication and ending 5 years thereafter. Proposals should be submitted to main investigator.
Supporting Information: Study Protocol, SAP, ICF